CLINICAL TRIAL: NCT02120924
Title: A Multicenter, Double-blind, Randomized, Parallel-group, Vehicle-Controlled Study to Evaluate the Safety and Clinical Equivalence of a Generic Azelaic Acid Gel, 15% and the Reference Listed Finacea® (Azelaic Acid) Gel, 15% in Patients With Moderate Facial Rosacea.
Brief Title: A Study to Evaluate the Safety and Clinical Study of Azelaic Acid Gel 15% in Patients With Moderate Facial Rosacea
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Actavis Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 13-1014
Record Dates: First submitted 2014-04-21; First posted 2014-04-23 (Estimated); Results first posted 2020-06-02 (Actual); Last update posted 2020-06-02 (Actual); Status verified 2020-05

CONDITIONS: Rosacea
Keywords: Moderate facial rosacea; Azelaic acid; Rosacea
MeSH Terms: conditions — Rosacea | interventions — azelaic acid; Drugs, Generic; Gels

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Finacea (Active Comparator): Finacea® (azelaic acid) Gel, 15% (Intendis)
  Interventions: Drug: Finacea
- Azelaic Acid (Experimental): Azelaic Acid, 15% topical gel (Watson Laboratories, Inc.)
  Interventions: Drug: Azelaic acid
- Vehicle Gel (Placebo Comparator): Gel Vehicle of the test product (Watson Laboratories, Inc.)
  Interventions: Drug: Vehicle

INTERVENTIONS:
Drug: Azelaic acid — Dosage form: Topical gel Dosage: Apply gel to the affected areas of the face twice daily for 12 weeks. The amount needed depends upon the size of the lesion site. Assure that enough is applied to adequately cover each lesion. Normally 0.5 g of gel is used on each 5 cm x 5 cm lesion site.
  Other Names: Generic
  Arms: Azelaic Acid
Drug: Vehicle — Dosage form: Topical gel Dosage: Apply gel to the affected areas of the face twice daily for 12 weeks. The amount needed depends upon the size of the lesion site. Assure that enough is applied to adequately cover each lesion. Normally 0.5 g of gel is used on each 5 cm x 5 cm lesion site.
  Other Names: Placebo
  Arms: Vehicle Gel
Drug: Finacea — Dosage form: Topical gel Dosage: Apply gel to the affected areas of the face twice daily for 12 weeks. The amount needed depends upon the size of the lesion site. Assure that enough is applied to adequately cover each lesion. Normally 0.5 g of gel is used on each 5 cm x 5 cm lesion site.
  Other Names: Finacea® (azelaic acid) Gel, 15% (Intendis)
  Arms: Finacea

SUMMARY:
The purpose of the study is to compare the safety and efficacy profiles of a generic Azelaic Acid Gel, 15% to the reference listed Finacea® (azelaic acid) Gel, 15% in the treatment of moderate facial rosacea.

DETAILED DESCRIPTION:
FINACEA® (azelaic acid) GEL, 15% contains azelaic acid, a naturally occurring saturated dicarboxylic acid that has proven anti-inflammatory effects, as well as anti-keratinizing and antimicrobial action, although its mechanism of action in rosacea is not well understood. This study will be conducted in compliance with the protocol, Good Clinical Practices (GCP) and the applicable regulatory requirement(s). Marketed by Intendis, Finacea® (azelaic acid) Gel, 15% is a safe and effective topical therapy used for the treatment of moderate facial rosacea. Watson Laboratories, Inc. has developed a generic formulation of azelaic acid 15% gel and the current study is designed to evaluate the safety and efficacy of this formulation.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or non-pregnant female ≥18 years-of-age with a clinical diagnosis of moderate facial rosacea.
* Patient must have at least eight and not more than fifty inflammatory facial lesions (i.e., papules/pustules) and ≤2 nodules on the face. For the purposes of study treatment and evaluation, these lesions should be limited to the facial treatment area including those present on the nose. Lesions involving the eyes, and scalp should be excluded from the count.
* Patients must have persistent erythema on the face with moderate (Definite redness, easily recognized) to Severe (Marked erythema; fiery red).
* Patients must have a mild to moderate score for telangiectasia on the face - Patients must have a definite clinical diagnosis of moderate facial rosacea as per the IGE
* Patient must be willing to minimize external factors that might trigger rosacea flare-ups (e.g., spicy foods, thermally hot foods and drinks, hot environments, prolonged sun exposure, strong winds and alcoholic beverages).
* Patient must be in general good health and free from any clinically significant disease other than rosacea, that might interfere with the study evaluations.
* Patient must be willing and able to understand and comply with the requirements of the study, apply the medication as instructed, return for the required treatment period visits, comply with therapy prohibitions, and be able to complete the study.
* Female Subjects of childbearing potential (excluding women who are surgicallysterilized or postmenopausal for at least 1 year), in addition to having a negative urine pregnancy test, must be willing to use an acceptable form of birth control during the study from the day of the first dose administration to 30 days after the last administration of study drug For the purpose of this study the following are considered acceptable methods of birth control: oral contraceptives, contraceptive patches, contraceptive implant, vaginal contraceptive, double barrier methods (e.g., condom and spermicide), contraceptive injection (Depo-provera®), intrauterine device (IUD), hormonal IUD (Mirena®) and abstinence with a documented second acceptable method of birth control, should the patient become sexually active. Patients on hormonal contraception must be stabilized on the same type for at least three months prior to enrollment in the study and must not change the hormonal contraception during the study. Patients who had used hormonal contraception and stopped must have stopped no less than three months prior to the study. A sterile sexual partner is NOT considered an adequate form of birth control.
* All male patients must agree to use accepted methods of birth control with their partners, from the day of the first dose administration to 30 days after the last administration of study drug. Abstinence is an acceptable method of birth control. Female partners should use an acceptable method of birth control as described in the above Item Number 10.
* Patients who use make-up must have used the same brands/types of make-up for a minimum period of 14 days prior to study entry and must agree to use the same make-up, brand/type, or frequency of use, throughout the study.

Exclusion Criteria:

* Pregnant or lactating or planning to become pregnant during the study period.
* Presence of any skin condition on the face that would interfere with the diagnosis or assessment of rosacea.
* Excessive facial hair (e.g. beards, sideburns, moustaches, etc.) that would interfere with diagnosis or assessment of rosacea.
* History of hypersensitivity or allergy to azelaic acid, propylene glycol or any other component of the formulation.
* The use within 6 months prior to baseline of oral retinoids (e.g. Accutane®) or therapeutic vitamin A supplements of greater than 10,000 units/day (multivitamins are allowed).
* The use of estrogens or oral contraceptives for less than 3 months prior to baseline.
* The use within 1 month prior to baseline of:

  1. topical retinoids to the face;
  2. systemic antibiotics known to have an impact on the severity of facial rosacea (e.g., containing tetracycline and its derivatives, erythromycin and its derivatives, sulfamethoxazole, or trimethoprim);
  3. systemic corticosteroids (Note: intranasal and inhalational corticosteroids do not require a washout and maybe used throughout the trial if the subject is on a stable dose).
* Use within 2 weeks prior to baseline of:

  1. topical corticosteroids;
  2. topical antibiotics;
  3. topical medications for rosacea (e.g., metronidazole).
* Patients with moderate or severe rhinophyma, dense telangiectases (score 3, severe), or plaque-like facial edema.
* Patients with a severe irritation grade for erythema, dryness, scaling, pruritus, stinging/burning, and edema.
* Ocular rosacea (e.g., conjunctivitis, blepharitis, or keratitis) of sufficient severity to require topical or systemic antibiotics.
* A patient who has used a sauna during the 2 weeks prior to study entry and during the study.
* Patients who have performed wax epilation of the face within 14 days prior to baseline
* A patient who has a history of being unresponsive to topical azelaic acid therapy.
* A patient with bacterial folliculitis.
* A patient who consumes excessive alcohol, abuses licit or illicit drugs, or has a condition that could compromise the patient's ability to comply with study requirements.
* Patients who engage in activities that involve excessive or prolonged exposure to sunlight or weather extremes, such as wind or cold.
* A patient who has any clinically significant condition or situation, other than the condition being studied that, in the opinion of the Investigator, would interfere with the study evaluations or optimal participation in the study.
* A patient who has used any topical azelaic acid therapy within 30 days of baseline visit.
* Patients who have participated in an investigational drug study (i.e., patients have been treated with an Investigational Drug) within 30 days prior to baseline will be excluded from study participation. Patients who are participating in non-treatment studies such as observational studies or registry studies can be considered for inclusion.
* Patients who have been previously enrolled in this study.
* Patients who have had laser therapy (for telangiectasia or other conditions), electrodessication and phototherapy (e.g., ClearLight®) to the facial area within 180 days prior to study entry.
* Patients who have had cosmetic procedures (e.g., facials) which may affect the efficacy and safety profile of the Investigational Product within 14 days prior to study entry.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1009 (Actual)
Dates: Start 2013-07; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Capicchioni, Study Director — Akesis, LLC
Locations (30):
- United States (30):
  - Site 24, Fremont, California
  - Site 22, Santa Monica, California
  - Site 1, Brandon, Florida
  - Site 3, Fort Myers, Florida
  - Site 27, Jacksonville, Florida
  - Site 19, Miami, Florida
  - Site 9, Miami, Florida
  - Site 29, Miramar, Florida
  - Site 2, Tampa, Florida
  - Site 15, Chicago, Illinois
  - Site 4, Plainfield, Indiana
  - Site 14, Lake Charles, Louisiana
  - Site 17, Glenn Dale, Maryland
  - Site 6, Bay City, Michigan
  - Site 30, Clinton Township, Michigan
  - Site 16, Las Vegas, Nevada
  - Site 11, Raleigh, North Carolina
  - Site 23, Winston-Salem, North Carolina
  - Site 26, Philadelphia, Pennsylvania
  - Site 12, Warwick, Rhode Island
  - Site 28, Simpsonville, South Carolina
  - Site 20, Nashville, Tennessee
  - Site 21, College Station, Texas
  - Site 5, Dallas, Texas
  - Site 8, El Paso, Texas
  - Site 13, Houston, Texas
  - Site 7, Katy, Texas
  - Site 18, Salt Lake City, Utah
  - Site 10, Norfolk, Virginia
  - Site 25, University Place, Virginia

RESULTS

PARTICIPANT FLOW:
Groups:
- Azelaic Acid, 15% Topical Gel: Test product: Azelaic Acid, 15% topical gel (Watson Laboratories, Inc.)
  Azelaic acid: Dosage form: Topical gel Dosage: Apply gel to the affected areas of the face twice daily for 12 weeks. The amount needed depends upon the size of the lesion site. Assure that enough is applied to adequately cover each lesion. Normally 0.5 g of gel is used on each 5 cm x 5 cm lesion site.
- Finacea® (Azelaic Acid) Gel, 15% (Intendis): Reference product: Finacea® (azelaic acid) Gel, 15% (Intendis)
  Azelaic acid: Dosage form: Topical gel Dosage: Apply gel to the affected areas of the face twice daily for 12 weeks. The amount needed depends upon the size of the lesion site. Assure that enough is applied to adequately cover each lesion. Normally 0.5 g of gel is used on each 5 cm x 5 cm lesion site.
- Gel Vehicle: Placebo product: Gel Vehicle of the test product (Watson Laboratories, Inc.)
  Azelaic acid: Dosage form: Topical gel Dosage: Apply gel to the affected areas of the face twice daily for 12 weeks. The amount needed depends upon the size of the lesion site. Assure that enough is applied to adequately cover each lesion. Normally 0.5 g of gel is used on each 5 cm x 5 cm lesion site.
Period: Overall Study
Arm/Group | Azelaic Acid, 15% Topical Gel | Finacea® (Azelaic Acid) Gel, 15% (Intendis) | Gel Vehicle
Started | 404 | 403 | 202
Completed | 362 | 357 | 173
Not Completed | 42 | 46 | 29
Not completed — Lack of Efficacy | 1 | 2 | 3
Not completed — Adverse Event | 0 | 1 | 3
Not completed — Withdrawal by Subject | 16 | 20 | 8
Not completed — Lost to Follow-up | 14 | 14 | 11
Not completed — Pregnancy | 2 | 0 | 0
Not completed — Protocol Violation | 3 | 7 | 2
Not completed — Physician Decision | 0 | 1 | 1
Not completed — Death | 1 | 0 | 0
Not completed — Compliance with IP | 5 | 1 | 1

BASELINE CHARACTERISTICS:
Population: Summary of Demographic characteristics in PP Population
Groups:
- Finacea® (Azelaic Acid) Gel, 15%: Reference product: Finacea® (azelaic acid) Gel, 15% (Intendis)
  Azelaic acid: Dosage form: Topical gel Dosage: Apply gel to the affected areas of the face twice daily for 12 weeks. The amount needed depends upon the size of the lesion site. Assure that enough is applied to adequately cover each lesion. Normally 0.5 g of gel is used on each 5 cm x 5 cm lesion site.
- Total: Total of all reporting groups
Arm/Group | Azelaic Acid, 15% Topical Gel | Finacea® (Azelaic Acid) Gel, 15% | Gel Vehicle | Total
Number analyzed (Participants) | 293 | 274 | 127 | 694
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.4 (12.71) | 50.0 (12.42) | 51.4 (11.73) | 50.8 (12.42)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 195 | 195 | 89 | 479
  Male | 98 | 79 | 38 | 215
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 118 | 126 | 59 | 303
  Not Hispanic or Latino | 175 | 148 | 68 | 391
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 3 | 2 | 1 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 0 | 1
  Black or African American | 0 | 0 | 0 | 0
  White | 280 | 263 | 124 | 667
  More than one race | 10 | 8 | 2 | 20
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline to Week 12 in the Inflammatory (Papules and Pustules) Lesion Counts.
Description: Percent change from baseline to Week 12 in the inflammatory (papules and pustules) lesion counts in PP population.
Time Frame: Baseline to Week 12
Population: Per protocol population
Measure: Mean (Standard Deviation); unit: Percent change in lesion counts
Groups:
- Gel Vehicle: Placebo product (Watson Laboratories, Inc.)
  Azelaic acid: Dosage form: Topical gel Dosage: Apply gel to the affected areas of the face twice daily for 12 weeks. The amount needed depends upon the size of the lesion site. Assure that enough is applied to adequately cover each lesion. Normally 0.5 g of gel is used on each 5 cm x 5 cm lesion site.
Arm/Group | Azelaic Acid, 15% Topical Gel | Finacea® (Azelaic Acid) Gel, 15% | Gel Vehicle
Number analyzed (Participants) | 293 | 274 | 127
Percent change in lesion counts | -66.96 (29.394) | -68.62 (27.415) | -38.64 (46.845)
Statistical Analysis 1: Comparison: Azelaic Acid, 15% Topical Gel vs Finacea® (Azelaic Acid) Gel, 15%; The primary endpoint was the percent change from baseline to Week 12 in the inflammatory (papules and pustules) lesion counts in PP population; Test type: Equivalence — Bioequivalence was established if the 90% CI for the ratio of Test/Reference means was contained within the interval [0.80, 1.25]; Mean Difference (Net) = 0.98, 90% CI 2-sided [0.92 to 1.05] — Bioequivalence was established if the 90% CI for the ratio of Test/Reference means was contained within the interval [0.80, 1.25]

2. Secondary Outcome: The Percentage of Subjects With a Clinical Response of "Success" at Week 12 Using Investigator Global Evaluation (IGE)
Description: The secondary endpoint is the clinical response of "success" or "failure" at Week 12 on the IGE. Success is defined as an IGE score of 0 (clear) or 1 (almost clear). Any subject who is not considered to be a success will be considered to be a failure.
  Score-Grade-Definition 0 - Clear - No inflammatory lesions present; at most, mild erythema.
  1. - Almost Clear - Very mild erythema present. Very few small papules/pustules.
  2. - Mild - Mild erythema. Several small papules/pustules.
  3. - Moderate - Moderate erythema. Several small or large papules/pustules, and up to two nodules.
  4. - Severe - Severe erythema. Numerous small and/or large papules/pustules, up to several nodules.
Time Frame: Baseline to 12 weeks
Population: Analysis of Treatment Success Based on IGE Score at Week 12 in PP Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Azelaic Acid, 15% Topical Gel | Finacea® (Azelaic Acid) Gel, 15% | Gel Vehicle
Number analyzed (Participants) | 293 | 274 | 127
Participants
  Success | 138 | 117 | 40
  Failure | 155 | 157 | 87
Statistical Analysis 1: Comparison: Azelaic Acid, 15% Topical Gel vs Finacea® (Azelaic Acid) Gel, 15%; Test type: Equivalence — A two-sided, continuity-corrected, 90% CI on the Test-to-Reference difference for the proportion of subjects with treatment success on the IGE was constructed; Mean Difference (Net) = 0.044, 90% CI 2-sided [-0.028 to 0.116] — Bioequivalence was established if the 90% CI for the difference was contained within the interval [-0.20, +0.20]

ADVERSE EVENTS:
Time Frame: Adverse events were monitored and collected over a period of at least 12 weeks, through to study completion.
Arm/Group | Azelaic Acid, 15% Topical Gel | Finacea® (Azelaic Acid) Gel, 15% | Gel Vehicle
All-Cause Mortality (participants affected / at risk) | 1/390 | 0/386 | 0/190
Serious Adverse Events (participants affected / at risk) | 1/390 | 0/386 | 0/190
Other Adverse Events (participants affected / at risk) | 109/390 | 98/386 | 47/190
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Azelaic Acid, 15% Topical Gel (N=390) | Finacea® (Azelaic Acid) Gel, 15% (N=386) | Gel Vehicle (N=190)
Cardiac failure congestive (Cardiac disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Azelaic Acid, 15% Topical Gel (N=390) | Finacea® (Azelaic Acid) Gel, 15% (N=386) | Gel Vehicle (N=190)
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 1 | 0 | 0
Ear pain (Ear and labyrinth disorders) | 1 | 0 | 1
Vertigo (Ear and labyrinth disorders) | 1 | 0 | 0
Hypothyroidism (Endocrine disorders) | 0 | 0 | 1
Blepharospasm (Eye disorders) | 1 | 0 | 0
Eye irritation (Eye disorders) | 1 | 0 | 0
Eye pain (Eye disorders) | 1 | 0 | 0
Eye pruritus (Eye disorders) | 0 | 1 | 0
Foreign body sensation in eye (Eye disorders) | 1 | 0 | 0
Lacrimation increased (Eye disorders) | 1 | 1 | 0
Vision blurred (Eye disorders) | 1 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 2
Abdominal pain (Gastrointestinal disorders) | 1 | 1 | 0
Abdominal pain lower (Gastrointestinal disorders) | 1 | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 3 | 3 | 0
Aphthous stomatitis (Gastrointestinal disorders) | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 2 | 5 | 2
Dyspepsia (Gastrointestinal disorders) | 1 | 5 | 0
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 | 1 | 1
Haemorrhoids (Gastrointestinal disorders) | 0 | 1 | 1
Mouth ulceration (Gastrointestinal disorders) | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 5 | 1 | 0
Tooth crowding (Gastrointestinal disorders) | 1 | 0 | 0
Toothache (Gastrointestinal disorders) | 0 | 2 | 1
Vomiting (Gastrointestinal disorders) | 1 | 4 | 0
Adverse drug reaction (General disorders) | 0 | 0 | 1
Application site pain (General disorders) | 2 | 1 | 1
Application site pruritus (General disorders) | 1 | 0 | 0
Chills (General disorders) | 0 | 1 | 1
Fatigue (General disorders) | 2 | 2 | 0
Feeling hot (General disorders) | 1 | 0 | 0
Influenza like illness (General disorders) | 0 | 3 | 1
Local swelling (General disorders) | 1 | 0 | 0
Malaise (General disorders) | 0 | 1 | 0
Pain (General disorders) | 2 | 3 | 1
Pyrexia (General disorders) | 2 | 0 | 0
Biliary colic (Hepatobiliary disorders) | 1 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 1 | 0 | 0
Hypersensitivity (Immune system disorders) | 1 | 0 | 1
Seasonal allergy (Immune system disorders) | 0 | 1 | 0
Acute sinusitis (Infections and infestations) | 1 | 0 | 0
Alveolar osteitis (Infections and infestations) | 0 | 1 | 0
Atypical pnuemonia (Infections and infestations) | 0 | 0 | 1
Bacterial infection (Infections and infestations) | 0 | 1 | 0
Bronchitis (Infections and infestations) | 0 | 3 | 1
Cellulitis (Infections and infestations) | 0 | 0 | 1
Conjunctivitis bacterial (Infections and infestations) | 1 | 0 | 0
Conjunctivitis infective (Infections and infestations) | 0 | 1 | 0
Ear infection (Infections and infestations) | 2 | 0 | 0
Eye infection (Infections and infestations) | 0 | 1 | 0
Fungal infection (Infections and infestations) | 0 | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 1 | 0
Gastroenteritis viral (Infections and infestations) | 0 | 3 | 0
Herpes simplex (Infections and infestations) | 0 | 1 | 0
Hordeolum (Infections and infestations) | 0 | 1 | 0
Influenza (Infections and infestations) | 6 | 4 | 1
Kidney infection (Infections and infestations) | 0 | 1 | 0
Lyme disease (Infections and infestations) | 0 | 0 | 1
Nasopharyngitis (Infections and infestations) | 27 | 19 | 9
Oral herpes (Infections and infestations) | 0 | 1 | 0
Pertussis (Infections and infestations) | 1 | 1 | 0
Pharyngitis (Infections and infestations) | 0 | 1 | 0
Pharyngitis streptococcal (Infections and infestations) | 1 | 0 | 0
Sinusitis (Infections and infestations) | 6 | 7 | 1
Skin infection (Infections and infestations) | 0 | 0 | 1
Subcutaneous abscess (Infections and infestations) | 1 | 0 | 0
Tonsillitus (Infections and infestations) | 0 | 1 | 0
Tooth abscess (Infections and infestations) | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 3 | 5 | 3
Urinary tract infection (Infections and infestations) | 0 | 1 | 0
Foot fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Foreign body (Injury, poisoning and procedural complications) | 1 | 0 | 0
Post procedural complication (Injury, poisoning and procedural complications) | 0 | 1 | 0
Spinal column injury (Injury, poisoning and procedural complications) | 1 | 0 | 0
Sunburn (Injury, poisoning and procedural complications) | 0 | 1 | 0
Blood cholesterol increased (Investigations) | 0 | 1 | 0
Heart rate increased (Investigations) | 0 | 1 | 0
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Vitamin D deficiency (Metabolism and nutrition disorders) | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 1 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 4 | 5 | 0
Invertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1 | 2
Muscoloskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Burning sensation (Nervous system disorders) | 4 | 5 | 0
Dizziness (Nervous system disorders) | 1 | 0 | 0
Dizziness exertional (Nervous system disorders) | 0 | 1 | 0
Headache (Nervous system disorders) | 23 | 23 | 11
Migraine (Nervous system disorders) | 3 | 2 | 3
Nerve compression (Nervous system disorders) | 0 | 1 | 0
Neuropathy peripheral (Nervous system disorders) | 0 | 1 | 0
Paraesthesia (Nervous system disorders) | 0 | 1 | 0
Sinus headache (Nervous system disorders) | 0 | 1 | 1
Tension headache (Nervous system disorders) | 0 | 1 | 0
Transient ischaemic attack (Nervous system disorders) | 1 | 0 | 0
Anxiety (Psychiatric disorders) | 1 | 1 | 0
Hypertonic bladder (Renal and urinary disorders) | 0 | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 1 | 0 | 0
Dysmenorrhoea (Reproductive system and breast disorders) | 6 | 2 | 2
Premenstrual headache (Reproductive system and breast disorders) | 0 | 1 | 0
Allergic sinusitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 | 5 | 0
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 3 | 2 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 3
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 5 | 2 | 0
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Acne (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Blister (Skin and subcutaneous tissue disorders) | 0 | 2 | 0
Dermal cyst (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 2 | 2 | 2
Erythema (Skin and subcutaneous tissue disorders) | 5 | 4 | 4
Pain of skin (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 6 | 3 | 2
Rash (Skin and subcutaneous tissue disorders) | 0 | 4 | 0
Rosacea (Skin and subcutaneous tissue disorders) | 0 | 0 | 4
Skin burning sensation (Skin and subcutaneous tissue disorders) | 1 | 2 | 0
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Skin irritation (Skin and subcutaneous tissue disorders) | 2 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The results of the study may be published or presented by the Investigator(s) after the review by, and in consultation and agreement with the Sponsor, and such that confidential or proprietary information is not disclosed.